CLINICAL TRIAL: NCT07073963
Title: Virtual Patient Groups for Sarcoidosis Associated Fatigue
Acronym: SupportSarc
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Clinical and Translational Science Collaborative of Northern Ohio (Unknown); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-565; K23MD017284 (NIH); UM1TR004528 (NIH)
Record Dates: First submitted 2025-07-17; First posted 2025-07-20 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Sarcoidosis; Fatigue; Depression; Anxiety; Mental Health
Keywords: mindfulness; support group; virtual
MeSH Terms: conditions — Sarcoidosis; Fatigue; Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 8 week Virtual Mindfulness Based Cognitive Therapy Group (Experimental): This group will meet with a certified Mindfulness Based Cognitive Therapy counselor one time a week to learn and practice mindfulness techniques as a means of addressing fatigue and mental health in sarcoidosis. This group will fill out diaries of their use of Mindfulness Based Cognitive Therapy techniques for the duration of the 8 week intervention and complete fatigue, depression, and anxiety surveys at time 0, 8 weeks, and 5 months.
  Interventions: Behavioral: Virtual Mindfulness Based Cognitive Therapy Group
- Monthly Virtual Sarcoidosis Support group (Active Comparator): This group will be invited to join an existing virtual sarcoidosis support group. They will participate in the group for the 5 months of the trial. They will complete fatigue, depression, and anxiety surveys at time 0, 8 weeks, and 5 months.
  Interventions: Behavioral: Virtual sarcoidosis support group

INTERVENTIONS:
Behavioral: Virtual Mindfulness Based Cognitive Therapy Group — Mindfulness-Based Cognitive Therapy (MBCT) is an 8-week, group-based psychological intervention that integrates principles of cognitive behavioral therapy (CBT) with training in mindfulness meditation. The intervention is designed to help participants develop greater awareness of thoughts, emotions, and bodily sensations, with the goal of preventing depressive relapse and reducing psychological distress. Each weekly session includes guided mindfulness practices (e.g., body scan, sitting meditation, mindful movement), group discussion, and cognitive-behavioral exercises focused on recognizing and disengaging from unhelpful thought patterns. Participants are assigned daily home practice using audio recordings and written materials. The MBCT intervention will be delivered over a video platform for this trial.
  Arms: 8 week Virtual Mindfulness Based Cognitive Therapy Group
Behavioral: Virtual sarcoidosis support group — Participants attend a once-monthly, virtual support group via secure video conferencing. Each session includes a brief didactic presentation on topics relevant to living with chronic illness (e.g., symptom management, coping strategies, navigating healthcare) followed by a facilitated group discussion. The discussion emphasizes peer support, shared experiences, and emotional processing in a safe, respectful environment. Groups are led by an experienced facilitator with experience in chronic illness care. No home practice is required.
  Arms: Monthly Virtual Sarcoidosis Support group

SUMMARY:
This research study is testing whether Mindfulness-Based Cognitive Therapy (MBCT) can help reduce fatigue in people with sarcoidosis. The study will also look at whether MBCT can improve symptoms of anxiety and depression.

Participants will be placed into one of two groups:

* One group will take part in an 8-week virtual MBCT program, attend weekly online sessions, keep a daily mindfulness journal, and complete surveys about fatigue, anxiety, and depression.
* The other group will join a virtual support group once a month for 6 months and complete the same surveys.

The goal is to see which approach is more helpful for improving fatigue and mental well-being in people with sarcoidosis.

DETAILED DESCRIPTION:
Fatigue is a common and debilitating symptom of sarcoidosis. There are currently no approved treatments for sarcoidosis associated fatigue. We are testing an MBCT intervention based on previous work showing improvement of sarcoidosis associated fatigue with a virtual MBCT intervention in the Netherlands.

Participants will be adults diagnosed with sarcoidosis per ATS criteria and experiencing significant fatigue (Fatigue Assessment Scale [FAS] score ≥22). Participants will be recruited through Cleveland Clinic and partnering sarcoidosis clinics. Recruitment includes both in-person and virtual strategies using electronic health record (EHR) screening, MyChart messages, clinician referrals, and self-referral through a recruitment letter. Interested patients will complete eligibility screening, including a virtual or in-person consent process, FAS assessment, and online screener survey.

Following enrollment, participants will be randomized 1:1 to either the MBCT intervention or control group (support group). The MBCT intervention consists of 8 weekly, virtual group sessions led by trained facilitators and includes guided mindfulness practices, cognitive exercises, and home practice assignments. The control group will participate in an existing monthly virtual sarcoidosis support group, which includes a brief educational presentation and group discussion.

Study outcomes will be collected using online surveys at three timepoints: baseline (prior to intervention), 8 weeks (immediately post-MBCT), and 5 months (3-month follow-up). Outcomes include fatigue (primary), quality of life, depression, and anxiety. Qualitative interviews will be conducted after the intervention to explore participant experiences with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Meets ATS criteria diagnosis for sarcoidosis (as determined by recruiting physician)
* Fatigue defined as FAS score ≥ 22
* Age ≥ 18 years old
* Ability to speak and read English
* Access to internet
* Capacity to consent

Exclusion Criteria:

* Current daily meditation practice
* Prior history of engaging in formal mindfulness-based interventions including: MBSR, MBCT, Acceptance and Commitment therapy, Dialectical Behavior Therapy
* Any condition that would prevent being a suitable candidate for the group intervention (as determined by online screening questionnaire and screening interview)
* Comorbid psychiatric illness or clinical features that would interfere with participant's ability to participate in or receive benefit from the MBCT-T intervention, including but not limited to: active suicidal ideation; current or recent history (in the last six months) of psychosis or mania; borderline, histrionic or narcissistic personality disorder; cognitive impairment; sensory disabilities; discomfort participating in a group-based intervention, drug use
* Lack of interest in study participation (assessed by online screening questionnaire).
* Lack of access to any form of online video access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue Assessment Scale | From enrollment to the end of the study period at 5 months
  validated 10 items fatigue questionnaire reported as an aggregate score

SECONDARY OUTCOMES:
Kings Sarcoidosis Questionnaire - General Health | From enrollment to end of study period at 5 months
  The KSQ General Health is a 10-item self-report survey reported as a single aggregate score which assesses quality of life in sarcoidosis.
Patient Health Questionnaire - 8 | From enrollment to end of study period at 5 months
  It is a self-reported measure of depressive symptom severity and consists of items consistent with criteria for DSM-based diagnosis. PHQ-8 scores range from 0 to 24. Each of the 8 items can be scored from 0 ("not at all") to 3 ("nearly every day"). Cut-points of 5, 10, 15, and 20 represent the thresholds for mild, moderate, moderately severe, and severe depression, respectively. The construct validity of the PHQ-8 has been demonstrated in a wide range of patient populations
Generalized Anxiety Disorder-7 | From enrollment to end of study period at 5 months
  7-item questionnaire that measures frequency of anxiety symptoms over the past 7 days. Response options are scored on a 4-point Likert scale ranging from "not at all" to "nearly every day." The summed score will be reported.

OTHER OUTCOMES:
Five Facet of Mindfulness Scale (Short Form; FFMQ-15) | From enrollment to end of study period at 5 months
  The FFMQ is a measure of treatment fidelity. The FFMQ measures pre-post trait mindfulness and is assessed using 15 items that index the degree to which participants experience daily mindfulness, a central objective of MBCT-V treatment. Each item is rated on a 5-point scale from '1' = never or very rarely true to '5' = very often or always true. Reported as a single aggregate score
Client Satisfaction Questionnaire (CSQ-8) | From enrollment to end of study period at 5 months
  The CSQ-8 is a validated questionnaire of patients satisfaction with mental health interventions. It involves summing response to 8 questions on a 4 point scale with scores ranging from 8 to 32.

CONTACTS AND LOCATIONS:
Overall Officials: Logan J Harper, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No